CLINICAL TRIAL: NCT04765137
Title: Targeting Cerebrovascular Reactivity for Precision Medicine: Pilot Trial of Atorvastatin
Brief Title: Evaluate the Effect of Atorvastatin on Cerebrovascular Reactivity in Mild Cognitive Impairment (MCI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Richman Family Precision Medicine Center of Excellence in Alzheimer Disease (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00256402
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Cerebral Vascular Reactivity
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Open-label study with atorvastatin 40 mg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atorvastatin 40 mg (Experimental): Participants receive 40 mg atorvastatin orally daily in the evening.
  Interventions: Drug: Atorvastatin Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin Oral Tablet — Atorvastatin pill 40 mg to be taken every night
  Other Names: Lipitor oral tablet

SUMMARY:
The purpose of this study is to evaluate the effect of atorvastatin on brain vessel reactivity and with it on blood flow in people with mild cognitive impairment.

DETAILED DESCRIPTION:
Participants are first being informed about potential benefits and risks of the study and are required to give written consent. After that participants will undergo detailed phone screen to determine eligibility for study entry. At week 0, participants who meet eligibility requirements will be prescribed atorvastatin (40 mg, once in the evening) in an open-label manner.

ELIGIBILITY:
Inclusion Criteria are chosen to include participants with MCI, enriched for vascular risk factors:

* MCI defined by Clinical Dementia Rating (CDR) of 0.5 or 1.0.
* Memory, processing speed, executive function, language - cognitive scores > 1.5 standard deviations below age-education norms.
* Not demented by history.
* Not taking statins currently or in the last 6 months.
* Cognitive/functional impairment not likely due to another neurological disease or delirium.

Exclusion Criteria:

* Taking a statin currently or have taken a statin in the last 6 months.
* Contraindications to taking a statin.
* Transplant patient taking cyclosporine.
* Unable to undergo MRI procedures (such as having an implanted pacemaker or defibrillator or stimulator or having non MRI compatible metal).
* Diagnosis of dementia by history.
* Current diagnosis of substance abuse.
* History of stroke or myocardial infarction in past 6 months.
* History of HIV.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of MRI whole brain cerebrovascular reactivity (wbCVR) | Baseline and 12 weeks
  MRI based CVR is a newer technique that measures dilatory function of the microvessels which have been shown to be superior to measurement of Cerebral blood flow (CBF) and have also been shown to be low in participants with MCI.

SECONDARY OUTCOMES:
Change in plasma exosomes | Baseline and 12 weeks
  Endothelial-derived exosomes (EDE) reflect the neurochemistry of cerebrovascular endothelial cells, while neuronal-enriched extracellular vesicles (nEV) are associated with brain white matter hyperintensities.
Change in cognitive function (global neurocognitive measure) | Baseline and 12 weeks
  Assessed by Global neurocognitive measure.
Change in cognitive function (domain-specific neurocognitive measure) | Baseline and 12 weeks
  Assessed by Domain-specific neurocognitive measure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rosenberg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No